CLINICAL TRIAL: NCT01117441
Title: International Collaborative Treatment Protocol For Children And Adolescents With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Martin Schrappe, Prof. Dr. med., University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: AIEOP-BFM ALL 2009
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — pegaspargase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; Etoposide; Ifosfamide; Mercaptopurine; Methotrexate; Prednisone; Thioguanine; Vincristine; Vindesine; fludarabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- R1 control arm (Active Comparator): see detailed protocol description
  Interventions: Drug: PEG-L-asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: Radiation Therapy
- R1 experimental arm (Experimental): see detailed protocol description
  Interventions: Drug: PEG-L-asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: Radiation Therapy
- R2 control arm (Active Comparator): see detailed protocol description
  Interventions: Drug: PEG-L-asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: Radiation Therapy
- R2 experimental arm (Experimental): see detailed protocol description
  Interventions: Drug: PEG-L-asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: Radiation Therapy
- R-HR control arm (Active Comparator): see detailed protocol description
  Interventions: Drug: PEG-L-asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Drug: vindesine; Drug: daunoxome; Drug: fludarabine; Radiation: Radiation Therapy
- R-HR experimental arm (Experimental): see detailed protocol description
  Interventions: Drug: PEG-L-asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Drug: vindesine; Drug: daunoxome; Drug: fludarabine; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: PEG-L-asparaginase — see detailed protocol description
  Other Names: Oncaspar medac
Drug: cyclophosphamide — see detailed protocol description
Drug: cytarabine — see detailed protocol description
Drug: daunorubicin hydrochloride — see detailed protocol description
Drug: dexamethasone — see detailed protocol description
Drug: doxorubicin hydrochloride — see detailed protocol description
Drug: etoposide — see detailed protocol description
  Arms: R-HR control arm; R-HR experimental arm
Drug: ifosfamide — see detailed protocol description
  Arms: R-HR control arm; R-HR experimental arm
Drug: mercaptopurine — see detailed protocol description
Drug: methotrexate — see detailed protocol description
Drug: prednisone — see detailed protocol description
Drug: thioguanine — see detailed protocol description
Drug: vincristine sulfate — see detailed protocol description
Drug: vindesine — see detailed protocol description
  Arms: R-HR control arm; R-HR experimental arm
Drug: daunoxome — see detailed protocol description; only given by patients with poor MRD-response during the high risk treatment
  Arms: R-HR control arm; R-HR experimental arm
Drug: fludarabine — see detailed protocol description; only given by patients with poor MRD-response during the high risk treatment
  Arms: R-HR control arm; R-HR experimental arm
Radiation: Radiation Therapy — for eligibility for radiotherapy see detailed protocol description

SUMMARY:
Rationale/Purpose: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating young patients with acute lymphoblastic leukemia (ALL).

This trial is studying several different combination chemotherapy regimens to compare how well they work in treating young patients with ALL.

Study objectives

Primary study questions:

* Non high-risk (non-HR) precursor-B ALL (pB-ALL) patients with TEL/AML1-negative ALL or unknown TEL/AML1 status and flow cytometry minimal residual disease (MRD) in bone marrow on day 15 <0.1% or with TEL/AML1-positive ALL (randomized study question R1): Can the daunorubicin dose in Protocol IA be safely reduced by 50 % with a non-inferior EFS and a reduction of toxicity (treatment-related mortality and AE/SAE in Protocol I)?
* Patients with pB-ALL and risk group medium risk (MR) (randomized study question R2): Can the clinical outcome be improved by protracted asparagine depletion achieved through application of intensified PEG-L-asparaginase during reintensification and early maintenance?
* High-risk (HR) patients (as identified by day 33 - randomized study question RHR): Can the clinical outcome be improved by protracted exposure to PEG-L-asparaginase during Protocol IB?

Secondary study questions:

* Standard risk (SR) patients identified by at least one sensitive marker: Is the clinical outcome comparable to that obtained in SR patients (identified with two sensitive markers) in AIEOP-BFM ALL 2000, or can the outcome even be improved with the use of PEG-L-asparaginase instead of native E. coli L-ASP?
* T-ALL non-HR patients: Can the high level of outcome which was obtained for these patients in study AIEOP-BFM ALL 2000 be preserved or even improved with the use of PEG-L-ASP instead of native E. coli L-ASP?
* HR patients with persisting high MRD levels despite the use of the HR blocks in the intensified consolidation phase "MRD Non-Responders": Is it possible to improve the outcome and to achieve a further reduction of leukemic cell burden by administration of an innovative treatment schedule (DNX-FLA)?
* Patients participating in the randomized asparaginase studies (pB-ALL/MR, HR): Are asparaginase activity and asparaginase antibodies associated with development of allergic reactions, and do they have an effect on the outcome of the patients?
* What is the relative value of different methods of MRD monitoring in the definition of alternative stratification systems within a BFM-oriented protocol?

DETAILED DESCRIPTION:
Risk Stratification

* T/non-HR: T-ALL in absence of any HR criteria (see below)
* pB/non-HR: pB-ALL in absence of any HR criteria (see below).

  * SR (polymerase chain reaction(PCR)-MRD-SR (MRD-negative on day 33 and 78) or, if no PCR-MRD result available, FCM d15 < 0.1%)
  * MR (no SR)
* HR: Prednisone poor-response (≥1000 blast cells/µl in peripheral blood on day 8), blast cells ≥10% in bone marrow on day 15 as measured by FCM, non-remission on day 33, positivity for MLL/AF4 or t(4;11), hypodiploidy (< 45 chromosomes), PCR-MRD-HR (MRD ≥10E-3 on day 78) or PCR-MRD-MR SER (only in pB-ALL, MRD ≥ 10-3 on day 33 and MRD positive at a level of < 10E-3 on day 78)

Chemotherapy

According to the risk group, patients receive the following chemotherapy elements:

T/non-HR: Protocol I, Protocol M, Protocol II and Maintenance pB/non-HR: Protocol I, Protocol M, Protocol II and Maintenance HR: Protocol I, HR-1', HR-2', HR-3', 3x Protocol III, Maintenance Patients of the HR group with PCR-MRD ≥10E-3 after element HR-3' are eligible for treatment with element DNX-FLA.

Protocol I Cytoreductive prephase: Prednisone (PDN) on days 1-7 and one dose of methotrexate (MTX) intrathecal (IT) on day 1 Protocol IA: Prednisone (PDN) on days 8 to 28 (21 days); vincristine (VCR) on days 8, 15, 22, 29 (4 doses); daunorubicin (DNR) on days 8, 15, 22 and 29 (4 doses); pegylated L-asparaginase (PEG-L-ASP) on days 12 and 26; MTX IT on days 12 and 33 and in case of blast cells in cerebrospinal fluid at diagnosis additional IT MTX is given on days 19 and 26.

Protocol IA': Only two doses of DNR on days 8 and 15 given to patients eligible for randomization R1 and randomized into the experimental arm Protocol IA-CPM: additional cyclophosphamide (CPM) on day 10 only in T-ALL patients with prednisone poor-response Protocol IA-Dexa (IAD): Dexamethasone (DXM) instead of PDN is given to all patients with T-ALL without any high-risk criteria as identified by day 8.

Protocol IB: CPM on days 36 and 64; cytarabine (ARA-C) on days 38-41, 45-48, 52-55 and 59-62; 6-mercaptopurine (6-MP) on days 36 to 63 (28 days); MTX IT on day 45 and 59 Protocol IB-ASP+: additional PEG-L-ASP on days 40, 47, 54, and 61 (4 doses) are given to the patients eligible for randomization RHR and randomized into the experimental arm.

Protocol M 6-MP on days 1- 56, high-dose MTX (HD-MTX) on days 8, 22, 36, 50 and MTX IT on days 8, 22, 36 and 50 Protocol II Protocol IIA: DXM on days 1 to 21 (21 days); VCR on days 8, 15, 22, 29 (4 doses); doxorubicine (DOX) on days 8, 15, 22 and 29 (4 doses); PEG-L-ASP on day 8 (1 dose); MTX IT on days 1 and 18 only in patients with initial CNS involvement.

Protocol IIA-ASP+: additional PEG-L-ASP on day 22 for patients eligible for randomization R2 and randomized into the experimental arm.

Protocol IIB: CPM on day 36; ARA-C on days 38-41 and 45-48; thioguanine (TG) on days 36 to 49 (14 days) and MTX IT on days 38 and 45.

Protocol IIB-ASP+: additional PEG-L-ASP on days 36 and 50 for eligible for randomization R2 and randomized into the experimental arm.

Protocol III DXM on days 1-15; VCR on days 1 and 8; DOX on days 1 and 8; PEG-L-ASP on day 1; CPM on day 15; ARA-C on days 17-20 and 24-27; TG on days 15 - 28 and MTX IT on days 17 and 24, also on day 1 in patients with initial CNS involvement HR-1' DXM on days 1-5; VCR on days 1 and 6; HD-MTX on day 1; CPM every 12 hours on days 2-4 (5 doses); HD-ARA-C every 12 hours on day 5 (2 doses); PEG-L-ASP on day 6, MTX IT on day 1 HR-2' DXM on days 1 to 5; VDS on days 1 and 6; HD-MTX on day 1; IFO every 12 hours on days 2-4 (5 doses); DNR on day 5; PEG-L-ASP on day 6; MTX IT on day 1 and 1 in patients with initial CNS involvement also day 5 HR-3' DXM on days 1-5; ARA-C 4 x on days 1-2 in 12 h intervals; etoposide (VP-16) every 12 hours on days 3-5 (5 doses); PEG-L-ASP on day 6; MTX IT on day 1 DNX-FLA Flucytosine (FLU) on days 1-5 (5 doses); HD-ARA-C on days 1 to 5 (5 doses); liposomal daunorubicin (DNX) on days 1, 3 and 5 (3 doses); MTX IT on day 1

Interim/Maintenance (until week 104):

6-MP p.o. daily; MTX p.o. once a week, doses adjusted to white blood cell count; PEG-L-ASP: every second week (6 doses), only for patients eligible for randomization R2 and randomized into the experimental arm; MTX IT every 6 weeks up to a total of 6 doses for the following subgroups (all CNS-negative):

* T-ALL (HR or non-HR) with < 2 years of age at start of maintenance,
* T-ALL, non-HR and initial WBC < 100 000/μl
* pB-ALL with PPR and/or FCM-MRD day 15 ≥ 10 % and/or PCR-MRDMR SER as only HR criteria

Radiotherapy Patients without CNS involvement and

* T-ALL/non-HR, WBC ≥ 100 000/μl, and age ≥ 2 years at start of pCRT or
* with risk group HR and age ≥ 2 years at start of pCRT except pB-ALL with PPR and/or FCM-MRD day 15 ≥ 10 % and/or PCR-MRD-MR SER as only HR criteria receive preventive cranial radiotherapy with 12 Gy

Patients with CNS involvement receive therapeutic cranial radiotherapy with 18 Gy (age 1 to <2 years 12 Gy).

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed acute lymphoblastic leukemia
* age ≥ 1 year (> 365 days) and < 18 years old (up to 17 years old and 365 days)
* no Ph+ (BCR/ABL or t(9;22)-positive) ALL
* no evidence of pregnancy or lactation period
* no participation in another clinical study
* patient enrolled in a participating center
* written informed consent

Exclusion Criteria:

* pre-treatment with cytostatic drugs
* pre-treatment with cytostatic drugs
* steroid pre-treatment with ≥ 1 mg/kg/d for more than two weeks during the last month before diagnosis
* treatment started according to another protocol
* underlying diseases that prohibit treatment according to the protocol
* ALL diagnosed as second malignancy steroid pre-treatment with ≥ 1 mg/kg/d for more than two weeks during the last month before diagnosis

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6136 (Actual)
Dates: Start 2010-06; Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 10 years from the start of recruitment
  * Randomization R1: Event-free survival from time of randomization
  * Historical comparison non-HR T-ALL: Event-free survival from diagnosis
  * Historical comparison "MRD Non-Responders": Event-free survival from start of DNX-FLA (morphological non-response after HR-3' is no event for this study question)
Disease-free survival | 10 years from the start of recruitment
  * Randomization R2: Disease-free survival from time of randomization
  * Historical comparison SR: Disease-free survival from start of Protocol M
minimal residual disease (MRD) | week 12 of treatment
  Randomization RHR: rate of MRD highly positive patients (MRD ≥ 10-3) at TP2 (week 12)

SECONDARY OUTCOMES:
survival | 10 years from the start of recruitment
  All randomized and historical comparisons: Survival
treatment-related mortality | up to 25 months from the diagnosis
  All randomized and historical comparisons: treatment-related mortality in induction or CCR (overall and by chemotherapy/SCT)
adverse events | up to 25 months from the diagnosis
  All randomized and historical comparisons: incidence and frequency of adverse events of interest and serious adverse events
event-free survival | 10 years from the start of recruitment
  Randomization R-HR: Event-free survival from time of randomization
minimal residual disease | after 24 weeks of treatment
  "MRD Non-Responders": MRD levels after DNX-FLA

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schrappe, MD PhD, Principal Investigator — Department of Pediatrics, University Hospital of Schleswig-Holstein, Campus Kiel
Locations (139):
- Australia (2):
  - The Sydney Children's Hospital, Centre for Children's Cancer and Blood Disorders, Randwick
  - The Children's Hospital at Westmead, Department of Oncology, Westmead
- Austria (8):
  - Krankenhaus Dornbirn, Abt. für Kinder- und Jugendheilkunde, Dornbirn
  - Univ.-Kinderklinik Graz, Abt. Pädiatrische Hämato-Onkologie, Graz
  - Department f. Kinder- u. Jugendheilkunde, Universitätsklinik f. Pädiatrie II, Innsbruck
  - A.oe. Landeskrankenhaus Klagenfurt, Abt. für Kinder- und Jugendheilkunde, Klagenfurt
  - A.oe. Landeskrankenhaus Leoben, Abt. für Kinder und Jugendliche, Leoben
  - Landes-Kinderklinik Linz, Haematologie/Onkologie, Linz
  - St. Johanns Spital / Landeskrankenhaus, Salzburg, Kinderspital Abt. Kinder u. Jugendheilkunde, Salzburg
  - St. Anna Kinderspital, Zentrum für Kinder- und Jugendheilkunde, Vienna
- Czechia (8):
  - University Hospital Brno, Department of Pediatric Oncology, Brno
  - Regional Hospital České Budějovice, Department of Pediatrics, České Budějovice
  - University Hospital Hradec Králové, Department of Pediatrics, Hradec Králové
  - University Hospital Olomouc, Department of Pediatrics, Olomouc
  - Teaching Hospital Ostrava-Poruba, Department of Pediatrics, Ostrava-Poruba
  - University Hospital Plzeň, Department of Pediatrics, Pilsen
  - University Hospital Motol, Department of Pediatric Hematology and Oncology, Prague
  - Masaryk´s Hospital Ústí nad Labem, Department of Pediatrics, Ústí nad Labem
- Germany (52):
  - Kinderklinik der med. Fakultät der RWTH, Bereich Hämatologie/Onkologie, Aachen
  - I. Klinik für Kinder u. Jugendliche, Klinikum Augsburg, Hämatologie/ Onkologie, Augsburg
  - Klinikum Bayreuth, Kinderklinik, Bayreuth
  - Klinikum Berlin-Buch II. Kinderklinik, Bereich Onkologie/Allg. Pädiatrie, Berlin
  - Kinderklinik der Charité, Campus Virchow Klinikum (CVK), Abt.: Kinderhämatologie, Berlin
  - Städtisches Krankenhaus, Kinderklinik, Braunschweig
  - Klinikum Chemnitz gGmbH, Klinik für Kinder- und Jugendmedizin, Hämatologie / Onkologie, Chemnitz
  - Kliniken der Stadt Köln GmbH, Kinderkrankenhaus Riehl, Cologne
  - Med. Einrichtungen der Universität zu Köln, Klinik für Allg. Kinderheilkunde, Onkologisch-hämatologische Station, Cologne
  - Carl-Thiem-Klinikum, Kinderklinik, Abt. Hämatologie/Onkologie, Cottbus
  - Vestische Kinder- u. Jugendklinik, Universitätsklinik Witten/Herdecke, Datteln
  - Klinikum Lippe-Detmold, Kinder- und Jugendmedizin, Detmold
  - Klinikum Dortmund, Klinik f. Kinder- und Jugendmedizin, Dortmund
  - Uni.Klinik Carl Gustav Carus, Klinik f. Kinderheilkunde, Dresden
  - Universitätskinderklinik, Düsseldorf
  - Helios Klinikum Erfurt GmbH, Klinik für Kinderheilkunde, Erfurt
  - Universitätsklinikum Erlangen, Kinder- und Jugendmedizin, Abt. für Onkologie/ Hämatologie/Immunologie, Erlangen
  - Universitätsklinikum Essen, Kinderklinik, Hämatologie/Onkologie, Essen
  - Universitäts-Kinderklinik, Klinik für Kinderheilkunde III, Pädiatrische Hämatologie/Onkologie, Frankfurt
  - Universitäts-Kinderklinik, Haematologie/ Onkologie, Freiburg im Breisgau
  - Klinikum der Justus-Liebig-Universität, Zentrum für Kinderheilkunde, Abt. Hämatologie/Onkologie, Giessen
  - Universitäts-Kinderklinik Päd. I, Hämatologie/Onkologie, Göttingen
  - Klinik und Poliklinik für Kinder und Jugendmedizin, Allgemeine Pädiatrie mit Poliklinik/Pädiatrische Onkologie und Hämatologie, Greifswald
  - Uniklinikum d. Martin Luther Universität, Halle Wittenberg, Univ.-und Poliklinik für Kinder- und Jugendmedizin, Halle
  - Medizinische Hochschule Hannover, Zentrum Kinderheilkunde u. Jugendmedizin, Hanover
  - Universitäts-Kinderklinik, Päd. Onkologie, Hämatologie, und Immunologie, Heidelberg
  - Klinikum Heilbronn GmbH, Klinik für Kinderheilkunde und Jugendmedizin/Perinatalzentrum, Heilbronn
  - Gemeinschaftskrankenhaus Herdecke, Kinderabteilung, Herdecke
  - Universitätsklinik für, Kinder- und Jugendmedizin, Päd. Hämatologie/ Onkologie, Homburg / Saar
  - Klinikum, der Friedrich-Schiller-Universität, Klinik für Kinder- und Jugendmedizin, Jena
  - Städtisches Klinikum Karlsruhe, Kinderklinik, Karlsruhe
  - Klinikum Kassel, Kinderklinik, Kassel
  - Klinik für Allgemeine Paediatrie, Univ.-Klinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Städtisches Krankenhaus Kemperhof, Kinderklinik, Koblenz
  - Department für Frauen- und Kindermedizin, Abteilung für Pädiatrische Onkologie, Hämatologie und Hämostaseologie, Leipzig
  - Universität zu Lübeck, Klinik für Kinder- u. Jugendmedizin, Abt. Hämatologie/ Onkologie/Immunologie, Lübeck
  - Universitätsklinikum Magdeburg, Klinik für Päd. Hämatologie/Onkologie, Magdeburg
  - Klinikum Mannheim gGmbH, Kinderklinik, Abt. Hämatologie/Onkologie, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Städt. Krankenhaus München GmbH, Krankenhaus München-Schwabingen, Kinderklinik d. TU, München
  - Universitäts-Kinderklinik, Päd. Hämatologie und Onkologie, Münster
  - Cnopf'sche Kinderklinik, Onkologie, Nuremberg
  - Klinikum Oldenburg gGmbH, Zentrum für Kinder- u. Jugendmedizin, (Elisabeth Kinderkrankenhaus), Oldenburg
  - Universitäts-Kinderklinik, Rostock
  - Asklepios-Klinik, Sankt Augustin GmbH, Sankt Augustin
  - HELIOS Kliniken Schwerin, Klinik f. Kinder-u. Jugendmedizin, Schwerin
  - Olga-Hospital, Kinderklinik, Pädiatrisches Zentrum, Abt. Hämatologie/Onkologie, Stuttgart
  - Krankenanstalt Trier, Mutterhaus der Borromaeerinnen, Pädiatrische Abteilung, Trier
  - Universitäts-Kinderklinik, Abt. Kinderheilkunde II, Hämatologie/Onkologie, Tübingen
  - Universitäts-Kinderklinik, Ulm
  - Stadtkrankenhaus, Kinderklinik, Wolfsburg
  - Universitäts-Kinderklinik, Würzburg
- Israel (8):
  - HaEmek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Bnai-Zion Medical Center, Haifa
  - Hadassah University Medical Center, Jerusalem
  - Schneider Children Medical Center of Israel, Petah Tikva
  - Dana children hospital, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (55):
  - Centro Regionale Oncoematologia Pediatrica Ospedale dei Bambini "G. Salesi" Clinica Pediatrica, Ancona
  - Dipartimento Biomedicina Età Evolutiva U.O Pediatrica I Policlinico, Bari
  - U.O.C. Pediatria e Patologia Neonatale Ospedale San Martino, Belluno
  - U.O. Pediatrica - OO.RR Bergamo, Bergamo
  - Istituto Ortopedico Rizzoli Sez. di chemioterapia dei tumori dell'apparato locomotore, Bologna
  - Oncologia ed Ematologia "Lalla Seràgnoli" Clinica Pediatrica Policlinico Sant'Orsola Malpighi, Bologna
  - Pediatria Ospedale Regionale, Bolzano
  - Clinica Pediatrica Oncoematologia pediatrica e TMO Ospedale dei Bambini, Brescia
  - Istituto di Clinica Pediatrica Ospedale Regionale per le Microcitemie, Cagliari
  - Divisione Ematologia - Oncologia Pediatrica Clinica Pediatrica, Catania
  - Unità Operativa di Ematologia ed Oncologia Pediatrica Az. Osp. "Pugliese-Ciaccio", Catanzaro
  - Unità Operativa Pediatria Azienda Ospedaliera Annuziata, Cosenza
  - Dipartimento di Medicina Clinica e Sperimentale Sezione di Pediatria Università di Ferrara, Ferrara
  - Dipartimento A.I. Oncoematologia Pediatrica e Cure Domiciliari U.O. Oncoematologia Pediatrica Azienda Ospedaliero-Universitaria Meyer, Florence
  - Dipartimento di Ematologia e Oncologia Pediatrica Instituto " G. Gaslini", Genova
  - Ospedale "Vito Fazzi" U.O. di Pediatria, Lecce
  - Clinica Pediatrica II De Marchi, Milan
  - Unità di Ricerca Clinica Pediatrica HSR TIGET - Istituto Scientifico San Raffaele, Milan
  - Divisione di Oncologia Pediatrica Ist. Nazionale Studio e Cura Tumori, Milan
  - Divisione Pediatria "Mariani" Ospedale "Niguarda Ca' Granda", Milan
  - U.O. di Ematologia, oncologia e trapianto Azienda Policlinico di Modena, Modena
  - Clinica Pediatrica dell'Università Milano - Bicocca A.O. San Gerardo - Fondazione MBBM, Monza
  - Dipartimento di Oncologia A.O. Santobono - Pausilipon, Napoli
  - A.O. "A. Cardarelli", U.O.S. Talassemia pediatrica ed emoglobinopatie pediatriche, Napoli
  - Servizio di Oncologia Pediatrica Dipartimento di Pediatria Seconda Università degli Studi di Napoli, Napoli
  - U.O.C. Pediatria - TIN, Ospedale "Umberto Primo" ASL SA - 1, Nocera Inferiore
  - S.C.D.U. Azienda Ospedaliera "Maggiore della carità", Novara
  - Dipartimento di Pediatria Università di Padova Cattedra Di Oncoematologia Pediatrica, Padua
  - Oncoematologia Pediatrica Ospedale dei Bambini G. di Cristina, Palermo
  - U.O. di Pediatria e Oncoematologia Pediatrica Az. Osp. Di Parma Ospedali Riuniti, Parma
  - Oncoematologia Pediatrica IRCCS, Policlinico San Matteo, Pavia
  - S.C. di Oncoematologia Pediatrica con Trapianto di CSE, Ospedale "S.M. della Misericordia" A.O. Perugia, Perugia
  - Ematologia, Ospedale di Muraglia, Pesaro
  - U.O. Pediatrica Azienda Ospedaliera San Salvatore, Pesaro
  - Dipartimento di Ematologia Ospedale Civile, Pescara
  - Centro di Oncoematologia Pediatrica e Trapianto Midollo Osseo Azienda Ospedaliero Universitaria Pisana Ospedale S. Chiara, Pisa
  - Centro Integrato di Emato-oncologia e dell'adolescenza A.O. S. Maria degli Angeli - Pordenone e IRCCS Centro di Riferimento Oncologico - Aviano, Pordenone
  - Divisione Ematologia Ospedali Riuniti, Reggio Calabria
  - U.O Pediatria Ospedale Infermi Azienda USL Rimini, Rimini
  - Ospedale Sant'Eugenio clinica pediatrica Univ. Tor Vergata, Roma
  - Oncoematologia pediatrica Università "La Sapienza" Roma, Roma
  - Sezione Ematologia Dipart. di biotecnologie Cellulari ed Ematologia Università "La Sapienza", Roma
  - Divisione di Ematologia Pediatrica Ospedale "Bambin Gesù"Istituto di Ricerca Scientifica, Roma
  - Divisione Oncologia Pediatrica Ospedale "Bambin Gesù", Roma
  - Divisione Oncologia Pediatrica Università Cattolica di Roma, Roma
  - U.O. Oncoematologia Pediatrica Ospedale "Casa Sollievo della Sofferenza", San Giovanni Rotondo
  - Clinica Pediatrica Università, Sassari
  - Dipartimento di Pediatria Ostetricia e Medicina della Riproduzione Università degli Studi di Siena, Siena
  - Ospedale Infantile Regina Margherita, Torino
  - Unità Operativa di Pediatria - U.T.I.N. Az.Osp. "Card. G. Panico", Tricase
  - U.O. Emato-Oncologia Pediatrica Università degli studi di Trieste Ospedale Infantile Burlo Garofolo, Trieste
  - SOS Oncologia Pediatrica Policlinico Universitario, Udine
  - Clinica Pediatrica Università degli Studi dell'Insubria di Varese Ospedale "Filippo del Ponte", Varese
  - U.O.C Oncoematologia Pediatrica Policlinico "G.B: Rossi", Verona
  - Ospedale San Bortolo, U.O. di Pediatria e patologia Neonatale, Vicenza
- Switzerland (6):
  - Kinderklinik, Hämatologie/Onkologie, Aarau
  - Baseler Kinderspital, Hämatologische Poliklinik, Basel
  - Repartio di Pediatria, Bellinzona
  - Pädiatrische Klinik, Kinderspital Luzern, Kinderonkologie, Lucerne
  - Hämatologie/Onkologie, Ostschweizer Kinderspital, FMH Pädiatrie, Hämatologie, Sankt Gallen
  - Kinderspital Zürich, Universitäts-Kinderklinik, Zurich

REFERENCES:
- [Background] Conter V, Bartram CR, Valsecchi MG, Schrauder A, Panzer-Grumayer R, Moricke A, Arico M, Zimmermann M, Mann G, De Rossi G, Stanulla M, Locatelli F, Basso G, Niggli F, Barisone E, Henze G, Ludwig WD, Haas OA, Cazzaniga G, Koehler R, Silvestri D, Bradtke J, Parasole R, Beier R, van Dongen JJ, Biondi A, Schrappe M. Molecular response to treatment redefines all prognostic factors in children and adolescents with B-cell precursor acute lymphoblastic leukemia: results in 3184 patients of the AIEOP-BFM ALL 2000 study. Blood. 2010 Apr 22;115(16):3206-14. doi: 10.1182/blood-2009-10-248146. Epub 2010 Feb 12. PMID 20154213
- [Background] Flohr T, Schrauder A, Cazzaniga G, Panzer-Grumayer R, van der Velden V, Fischer S, Stanulla M, Basso G, Niggli FK, Schafer BW, Sutton R, Koehler R, Zimmermann M, Valsecchi MG, Gadner H, Masera G, Schrappe M, van Dongen JJ, Biondi A, Bartram CR; International BFM Study Group (I-BFM-SG). Minimal residual disease-directed risk stratification using real-time quantitative PCR analysis of immunoglobulin and T-cell receptor gene rearrangements in the international multicenter trial AIEOP-BFM ALL 2000 for childhood acute lymphoblastic leukemia. Leukemia. 2008 Apr;22(4):771-82. doi: 10.1038/leu.2008.5. Epub 2008 Jan 31. PMID 18239620
- [Background] Moricke A, Zimmermann M, Reiter A, Henze G, Schrauder A, Gadner H, Ludwig WD, Ritter J, Harbott J, Mann G, Klingebiel T, Zintl F, Niemeyer C, Kremens B, Niggli F, Niethammer D, Welte K, Stanulla M, Odenwald E, Riehm H, Schrappe M. Long-term results of five consecutive trials in childhood acute lymphoblastic leukemia performed by the ALL-BFM study group from 1981 to 2000. Leukemia. 2010 Feb;24(2):265-84. doi: 10.1038/leu.2009.257. Epub 2009 Dec 10. PMID 20010625
- [Derived] Gottschalk H, Moricke A, Conter V, Schrappe M, Stary J, Cario G, Dworzak M, Attarbaschi A, Barbaric D, Locatelli F, Bodmer N, Elitzur S, Silvestri D, Dalla-Pozza L, Bergmann AK, Flotho C, Buldini B, Stanulla M, Izraeli S, Rizzari C, Bourquin JP, Biondi A, Valsecchi MG, Zimmermann M. Reducing Daunorubicin in Induction Therapy in Children With B-Lineage ALL With Favorable Prognosis: Results of Phase III Trial AIEOP-BFM ALL 2009. J Clin Oncol. 2025 Dec 10;43(35):3739-3749. doi: 10.1200/JCO-25-01357. Epub 2025 Nov 10. PMID 41213101
- [Derived] Conter V, Valsecchi MG, Cario G, Zimmermann M, Attarbaschi A, Stary J, Niggli F, Dalla Pozza L, Elitzur S, Silvestri D, Locatelli F, Moricke A, Engstler G, Smisek P, Bodmer N, Barbaric D, Izraeli S, Rizzari C, Boos J, Buldini B, Zucchetti M, von Stackelberg A, Matteo C, Lehrnbecher T, Lanvers-Kaminsky C, Cazzaniga G, Gruhn B, Biondi A, Schrappe M. Four Additional Doses of PEG-L-Asparaginase During the Consolidation Phase in the AIEOP-BFM ALL 2009 Protocol Do Not Improve Outcome and Increase Toxicity in High-Risk ALL: Results of a Randomized Study. J Clin Oncol. 2024 Mar 10;42(8):915-926. doi: 10.1200/JCO.23.01388. Epub 2023 Dec 14. PMID 38096462
- [Derived] Heilmann J, Vieth S, Moricke A, Attarbaschi A, Barbaric D, Bodmer N, Colombini A, Dalla-Pozza L, Elitzur S, Izraeli S, Mann G, Niggli F, Silvestri D, Stary J, Rizzari C, Valsecchi MG, Zapotocka E, Zimmermann M, Cario G, Schrappe M, Conter V. Effect of two additional doses of intrathecal methotrexate during induction therapy on serious infectious toxicity in pediatric patients with acute lymphoblastic leukemia. Haematologica. 2023 Dec 1;108(12):3278-3286. doi: 10.3324/haematol.2022.281788. PMID 37021527
- [Derived] Wurthwein G, Lanvers-Kaminsky C, Siebel C, Gerss J, Moricke A, Zimmermann M, Stary J, Smisek P, Schrappe M, Rizzari C, Zucchetti M, Hempel G, Wicha SG, Boos J; AIEOP-BFM ALL 2009 Asparaginase Working Party. Population Pharmacokinetics of PEGylated Asparaginase in Children with Acute Lymphoblastic Leukemia: Treatment Phase Dependency and Predictivity in Case of Missing Data. Eur J Drug Metab Pharmacokinet. 2021 Mar;46(2):289-300. doi: 10.1007/s13318-021-00670-8. Epub 2021 Feb 17. PMID 33595793
- [Derived] Tasian SK, Peters C. Targeted therapy or transplantation for paediatric ABL-class Ph-like acute lymphocytic leukaemia? Lancet Haematol. 2020 Dec;7(12):e858-e859. doi: 10.1016/S2352-3026(20)30369-0. No abstract available. PMID 33242441
- [Derived] Cario G, Leoni V, Conter V, Attarbaschi A, Zaliova M, Sramkova L, Cazzaniga G, Fazio G, Sutton R, Elitzur S, Izraeli S, Lauten M, Locatelli F, Basso G, Buldini B, Bergmann AK, Lentes J, Steinemann D, Gohring G, Schlegelberger B, Haas OA, Schewe D, Buchmann S, Moericke A, White D, Revesz T, Stanulla M, Mann G, Bodmer N, Arad-Cohen N, Zuna J, Valsecchi MG, Zimmermann M, Schrappe M, Biondi A. Relapses and treatment-related events contributed equally to poor prognosis in children with ABL-class fusion positive B-cell acute lymphoblastic leukemia treated according to AIEOP-BFM protocols. Haematologica. 2020 Jul;105(7):1887-1894. doi: 10.3324/haematol.2019.231720. Epub 2019 Oct 10. PMID 31601692
- [Derived] Kroll M, Kaupat-Bleckmann K, Morickel A, Altenl J, Schewel DM, Stanullal M, Zimmermann M, Schrappe M, Cario G. Methotrexate-associated toxicity in children with Down syndrome and acute lymphoblastic leukemia during consolidation therapy with high dose methotrexate according to ALL-BFM treatment regimen. Haematologica. 2020 Apr;105(4):1013-1020. doi: 10.3324/haematol.2019.224774. Epub 2019 Aug 1. PMID 31371414
- [Derived] Wurthwein G, Lanvers-Kaminsky C, Hempel G, Gastine S, Moricke A, Schrappe M, Karlsson MO, Boos J. Population Pharmacokinetics to Model the Time-Varying Clearance of the PEGylated Asparaginase Oncaspar(R) in Children with Acute Lymphoblastic Leukemia. Eur J Drug Metab Pharmacokinet. 2017 Dec;42(6):955-963. doi: 10.1007/s13318-017-0410-5. PMID 28349335